CLINICAL TRIAL: NCT01317147
Title: The Effect of Gastric Bypass on the Pharmacokinetics of Serotonin Reuptake Inhibitors
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: American Society for Metabolic and Bariatric Surgery (Other)
Responsible Party: Giselle Hamad, MD Assistant Professor of Surgery, University of Pittsburgh School of Medicine
Other Study IDs: PRO07120162
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Gastric Bypass; Depression; Anxiety Disorder
Keywords: pharmacokinetics; serotonin reuptake inhibitors; gastric bypass; depression; bioavailability; drug absorption; area under curve
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric bypass patients
  Interventions: Procedure: Roux-en-Y gastric bypass (RYGBP)

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass (RYGBP)

SUMMARY:
The morbidly obese frequently present with mood and anxiety disorders, which are often treated with serotonin reuptake inhibitors (SRI) antidepressant drugs. The investigators hypothesized that gastric bypass surgery would decrease the absorption of SRI. The investigators also wished to determine whether a reduction in SRI levels would increase the likelihood of worsening depressive symptoms.

DETAILED DESCRIPTION:
Twelve RYGB candidates who were successfully treated with an SRI for primary mood or anxiety disorders were studied prospectively. Blood samples for SRI plasma levels were drawn immediately after dose for pharmacokinetic studies (PK) preoperatively. Maximum concentration (CMAX), time to CMAX (TMAX), and Area Under Concentration/Time curve (AUC) were determined. PK studies were repeated at one, six, and twelve months post-operatively. PK data were corrected for dose at each study time point. The Structured Interview Guide for the Hamilton Depression Rating Scale- Atypical Depression Symptom Version was used to quantify depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerate general anesthesia
* Able to document prior unsuccessful attempts at weight loss under medical supervision during the last 6 months
* Able to provide informed consent
* Cleared for surgery by primary care MD, dietician, and psychiatrist
* SRI treatment specifically for depression for ≥6 wks at constant dose for last 2 out of 6 wks

Exclusion Criteria:

* pregnancy
* Unwilling or unable to comply with postoperative requirements for diet, supplements, exercise, or followup

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bariatric surgery clinic- Morbidly obese patients seeking RYGB who met criteria for bariatric surgery (BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with severe obesity-related comorbidities) and were received maintenance treatment with an SRI for primary mood or anxiety disorder.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-08; Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Hamad, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Onyike CU, Crum RM, Lee HB, Lyketsos CG, Eaton WW. Is obesity associated with major depression? Results from the Third National Health and Nutrition Examination Survey. Am J Epidemiol. 2003 Dec 15;158(12):1139-47. doi: 10.1093/aje/kwg275. PMID 14652298
- [Background] Sarwer DB, Cohn NI, Gibbons LM, Magee L, Crerand CE, Raper SE, Rosato EF, Williams NN, Wadden TA. Psychiatric diagnoses and psychiatric treatment among bariatric surgery candidates. Obes Surg. 2004 Oct;14(9):1148-56. doi: 10.1381/0960892042386922. PMID 15527626
- [Background] Alciati A, D'Ambrosio A, Foschi D, Corsi F, Mellado C, Angst J. Bipolar spectrum disorders in severely obese patients seeking surgical treatment. J Affect Disord. 2007 Aug;101(1-3):131-8. doi: 10.1016/j.jad.2006.11.008. Epub 2007 Jan 16. PMID 17229468
- [Background] Ali MR, Rasmussen JJ, Monash JB, Fuller WD. Depression is associated with increased severity of co-morbidities in bariatric surgical candidates. Surg Obes Relat Dis. 2009 Sep-Oct;5(5):559-64. doi: 10.1016/j.soard.2008.10.015. Epub 2008 Nov 21. PMID 19342306
- [Background] Serretti A, Mandelli L. Antidepressants and body weight: a comprehensive review and meta-analysis. J Clin Psychiatry. 2010 Oct;71(10):1259-72. doi: 10.4088/JCP.09r05346blu. PMID 21062615
- [Background] Malinowski SS. Nutritional and metabolic complications of bariatric surgery. Am J Med Sci. 2006 Apr;331(4):219-25. doi: 10.1097/00000441-200604000-00009. PMID 16617238
- [Background] Miller AD, Smith KM. Medication and nutrient administration considerations after bariatric surgery. Am J Health Syst Pharm. 2006 Oct 1;63(19):1852-7. doi: 10.2146/ajhp060033. PMID 16990631
- [Background] Pihlajamaki J, Gronlund S, Simonen M, Kakela P, Moilanen L, Paakkonen M, Pirinen E, Kolehmainen M, Karja V, Kainulainen S, Uusitupa M, Alhava E, Miettinen TA, Gylling H. Cholesterol absorption decreases after Roux-en-Y gastric bypass but not after gastric banding. Metabolism. 2010 Jun;59(6):866-72. doi: 10.1016/j.metabol.2009.10.004. Epub 2009 Dec 16. PMID 20015521
- [Background] Ruz M, Carrasco F, Rojas P, Codoceo J, Inostroza J, Rebolledo A, Basfi-fer K, Csendes A, Papapietro K, Pizarro F, Olivares M, Sian L, Westcott JL, Hambidge KM, Krebs NF. Iron absorption and iron status are reduced after Roux-en-Y gastric bypass. Am J Clin Nutr. 2009 Sep;90(3):527-32. doi: 10.3945/ajcn.2009.27699. Epub 2009 Jul 22. PMID 19625680
- [Background] Roerig JL, Steffen K, Zimmerman C, Mitchell JE, Crosby RD, Cao L. Preliminary comparison of sertraline levels in postbariatric surgery patients versus matched nonsurgical cohort. Surg Obes Relat Dis. 2012 Jan-Feb;8(1):62-6. doi: 10.1016/j.soard.2010.12.003. Epub 2010 Dec 15. PMID 21256091
- [Background] Skottheim IB, Stormark K, Christensen H, Jakobsen GS, Hjelmesaeth J, Jenssen T, Reubsaet JL, Sandbu R, Asberg A. Significantly altered systemic exposure to atorvastatin acid following gastric bypass surgery in morbidly obese patients. Clin Pharmacol Ther. 2009 Sep;86(3):311-8. doi: 10.1038/clpt.2009.82. Epub 2009 Jun 3. PMID 19494810
- [Background] Brolin RE. Update: NIH consensus conference. Gastrointestinal surgery for severe obesity. Nutrition. 1996 Jun;12(6):403-4. doi: 10.1016/s0899-9007(96)00154-2. PMID 8875533
- [Background] First MB, Spitzer RL, Gibbon M, Williams JBW. Structured clinical interview for DSM-IV axis I disorders-patient edition. : New York State Psychiatric Institute; 1996.
- [Background] Williams JBW, Terman M. Structured Interview Guide for the Hamilton Depression Rating Scale with Ayptical Depression Supplement (SIGH-ADS). New York: New York State Psychiatric Institute; 2003.
- [Background] Schauer PR, Ikramuddin S, Gourash W, Ramanathan R, Luketich J. Outcomes after laparoscopic Roux-en-Y gastric bypass for morbid obesity. Ann Surg. 2000 Oct;232(4):515-29. doi: 10.1097/00000658-200010000-00007. PMID 10998650
- [Background] Gubbins PO, Bertch KE. Drug absorption in gastrointestinal disease and surgery. Clinical pharmacokinetic and therapeutic implications. Clin Pharmacokinet. 1991 Dec;21(6):431-47. doi: 10.2165/00003088-199121060-00004. PMID 1782738
- [Background] Padwal R, Brocks D, Sharma AM. A systematic review of drug absorption following bariatric surgery and its theoretical implications. Obes Rev. 2010 Jan;11(1):41-50. doi: 10.1111/j.1467-789X.2009.00614.x. Epub 2009 Jun 2. PMID 19493300
- [Background] Magee SR, Shih G, Hume A. Malabsorption of oral antibiotics in pregnancy after gastric bypass surgery. J Am Board Fam Med. 2007 May-Jun;20(3):310-3. doi: 10.3122/jabfm.2007.03.060177. PMID 17478665
- [Background] Wills SM, Zekman R, Bestul D, Kuwajerwala N, Decker D. Tamoxifen malabsorption after Roux-en-Y gastric bypass surgery: case series and review of the literature. Pharmacotherapy. 2010 Feb;30(2):217. doi: 10.1592/phco.30.2.217. PMID 20099995
- [Background] Behrns KE, Smith CD, Sarr MG. Prospective evaluation of gastric acid secretion and cobalamin absorption following gastric bypass for clinically severe obesity. Dig Dis Sci. 1994 Feb;39(2):315-20. doi: 10.1007/BF02090203. PMID 8313814
- [Background] Seaman JS, Bowers SP, Dixon P, Schindler L. Dissolution of common psychiatric medications in a Roux-en-Y gastric bypass model. Psychosomatics. 2005 May-Jun;46(3):250-3. doi: 10.1176/appi.psy.46.3.250. PMID 15883146
- [Background] Brandacher G, Winkler C, Aigner F, Schwelberger H, Schroecksnadel K, Margreiter R, Fuchs D, Weiss HG. Bariatric surgery cannot prevent tryptophan depletion due to chronic immune activation in morbidly obese patients. Obes Surg. 2006 May;16(5):541-8. doi: 10.1381/096089206776945066. PMID 16687019
- [Background] Bodnar LM, Wisner KL. Nutrition and depression: implications for improving mental health among childbearing-aged women. Biol Psychiatry. 2005 Nov 1;58(9):679-85. doi: 10.1016/j.biopsych.2005.05.009. Epub 2005 Jul 25. PMID 16040007
- [Background] Hanley MJ, Abernethy DR, Greenblatt DJ. Effect of obesity on the pharmacokinetics of drugs in humans. Clin Pharmacokinet. 2010;49(2):71-87. doi: 10.2165/11318100-000000000-00000. PMID 20067334
- [Background] Kinzl JF, Schrattenecker M, Traweger C, Mattesich M, Fiala M, Biebl W. Psychosocial predictors of weight loss after bariatric surgery. Obes Surg. 2006 Dec;16(12):1609-14. doi: 10.1381/096089206779319301. PMID 17217637
- [Background] Legenbauer T, De Zwaan M, Benecke A, Muhlhans B, Petrak F, Herpertz S. Depression and anxiety: their predictive function for weight loss in obese individuals. Obes Facts. 2009;2(4):227-34. doi: 10.1159/000226278. Epub 2009 Aug 17. PMID 20054228
- [Background] Clark MM, Niaura R, King TK, Pera V. Depression, smoking, activity level, and health status: pretreatment predictors of attrition in obesity treatment. Addict Behav. 1996 Jul-Aug;21(4):509-13. doi: 10.1016/0306-4603(95)00081-x. PMID 8830908
- [Background] Rusch MD, Andris D. Maladaptive eating patterns after weight-loss surgery. Nutr Clin Pract. 2007 Feb;22(1):41-9. doi: 10.1177/011542650702200141. PMID 17242453
- [Background] Sanchez-Santos R, Del Barrio MJ, Gonzalez C, Madico C, Terrado I, Gordillo ML, Pujol J, Moreno P, Masdevall C. Long-term health-related quality of life following gastric bypass: influence of depression. Obes Surg. 2006 May;16(5):580-5. doi: 10.1381/096089206776945084. PMID 16687025
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Reis M, Aberg-Wistedt A, Agren H, Akerblad AC, Bengtsson F. Compliance with SSRI medication during 6 months of treatment for major depression: an evaluation by determination of repeated serum drug concentrations. J Affect Disord. 2004 Nov 1;82(3):443-6. doi: 10.1016/j.jad.2004.02.003. PMID 15555696